CLINICAL TRIAL: NCT06700395
Title: Phase I Clinical Study Evaluating the Tolerability and Pharmacokinetics of TQB2029 for Injection in Subjects With Multiple Myeloma
Brief Title: A Clinical Study of TQB2029 for Injection in Subjects With Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2029-I-01
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2029 injection (Experimental): TQB2029 injection, 28 days as a treatment cycle.
  Interventions: Drug: TQB2029 injection

INTERVENTIONS:
Drug: TQB2029 injection — TQB2029 for injection is a bispecific antibody targeting G Protein-Coupled Receptor, Class C, Group 5, Member D (GPRC5D) and Cluster of Differentiation 3 (CD3) . By recruiting and activating CD3 positive T cells, it induces T cells to kill malignant plasma cells expressing GPRC5D, thereby inhibiting the occurrence and development of tumors.

SUMMARY:
This is a study to evaluate the maximum tolerated dose (MTD), dose limiting toxicity (DLT), occurrence of all adverse events (AEs) and serious adverse events (SAEs), pharmacokinetic parameters, pharmacodynamic parameters, immunogenicity, and anti-tumor effects of TQB2029 for injection in Chinese adult subjects with multiple myeloma. The study is divided into Phase Ia and Ib, Phase Ia: dose escalation phase, to evaluate the safety and tolerability of TQB2029 for injection, and determining DLT and MTD; Phase Ib: Dose extension phase, to evaluate the effectiveness of TQB2029 for injection in subjects with multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who voluntarily join the study, sign the informed consent form, and have good compliance.
* Aged from 18 to 75 years; Eastern Cooperative Oncology Group performance status score: 0-2; at least 12 weeks expected survival period.
* Multiple myeloma with diagnostic records and meeting the International Myeloma Working Group (IMWG) diagnostic criteria
* There are measurable lesions present
* The function of main organs is normal.
* Subjects need to adopt effective methods of contraception.

Exclusion Criteria:

* Subjects who have taken Chinese patent medicines with anti-tumor indications in the drug instructions that National Medical Products Administration approved within 2 weeks before the first administration.
* Subjects who received targeted therapy or immunotherapy within 3 weeks before the first medication
* Subjects who is known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
* Subjects who has had or currently has other malignant tumors within the past 3 years prior to the first use of medication
* Subjects who with unrelieved toxic reactions above Common Terminology Criteria for Adverse Events (CTC AE) grade 1 caused by any previous treatment
* Subjects who have undergone major surgical treatment, significant traumatic injury, or are expected to undergo major surgery during the expected study treatment period within 4 weeks prior to the first use of medication
* Subjects who have experienced arterial/venous thrombotic event occurred within 6 months prior to the first administration
* Subjects with a history of psychotropic drug abuse unable to quit or with mental disorders;
* Subjects with any severe and/or uncontrolled disease
* According to the judgment of the investigators, there are accompanying diseases that seriously endanger the safety of patients or affect the completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2024-11-28 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) | During the first 28 days
  DLT refers to any of the following events in the first administration of TQB2029 for injection to the end of the first treatment cycle (C1D28) that the investigator and the sponsor consider to be related to the treatment of TQB2029 for injection.
Maximum tolerated dose (MTD) | Up to 18 months
  After the experiment is completed, sequential regression is used to determine the maximum tolerated dose (MTD). Specifically, calculate the toxicity rate of each dose group and select the dose closest to the target toxicity rate as MTD.
Recommended Phase II Dose (RP2D) | Up to 18 months
  Determine RP2D based on target toxicity rates for each dose group
Number of patients with adverse events (AEs) and serious adverse events (SAEs) | Up to 18 months
  Assessed by the National Cancer Institute Common Terminology Criteria for adverse events (NCI-CTCAE) v5.0.

SECONDARY OUTCOMES:
Elimination half-life (to be used in one-or non- compartmental model) (t1/2) | The first and second treatment cycle: 0 hours, 2 hours, 6 hours, 24 hours, 48 hours, 72 hours, 96 hours, 120 hours, 168 hours after dosing on the first day, 0 hours on the 15th day, and 0 hours on the 22nd day.
  t1/2 is time it takes for the blood concentration of TQB2029 or metabolite(s) to drop by half.
Maximum (peak) plasma drug concentration (Cmax) | The first and second treatment cycle: 0 hours, 2 hours, 6 hours, 24 hours, 48 hours, 72 hours, 96 hours, 120 hours, 168 hours after dosing on the first day, 0 hours on the 15th day, and 0 hours on the 22nd day.
  Cmax is the maximum plasma concentration of TQB2029 or metabolite(s).
Area under the plasma concentration-time curve from time zero to time t (AUC0-t) | The first and second treatment cycle: 0 hours, 2 hours, 6 hours, 24 hours, 48 hours, 72 hours, 96 hours, 120 hours, 168 hours after dosing on the first day, 0 hours on the 15th day, and 0 hours on the 22nd day.
  To characterize the pharmacokinetics of TQB2029 by assessment of area under the plasma concentration time curve from the first dose to infinity.
Apparent clearance rate (CL/F) | The first and second treatment cycle: 0 hours, 2 hours, 6 hours, 24 hours, 48 hours, 72 hours, 96 hours, 120 hours, 168 hours after dosing on the first day, 0 hours on the 15th day, and 0 hours on the 22nd day.
  The apparent clearance rate is used to predict dynamic distribution rates and evaluate the dynamics of nutrients.
Volume of distribution(Vz/F) | The first and second treatment cycle: 0 hours, 2 hours, 6 hours, 24 hours, 48 hours, 72 hours, 96 hours, 120 hours, 168 hours after dosing on the first day, 0 hours on the 15th day, and 0 hours on the 22nd day.
  Refers to the volume of bodily fluids required for drugs to be distributed in the body according to the plasma drug concentration at the time when the drug reaches dynamic equilibrium in the body.
Blood drug trough concentration (Cmin) | The first and second treatment cycle: 0 hours, 2 hours, 6 hours, 24 hours, 48 hours, 72 hours, 96 hours, 120 hours, 168 hours after dosing on the first day, 0 hours on the 15th day, and 0 hours on the 22nd day.
  Describe the minimum value of drug concentration.
Exploring the correlation between changes in cytokine levels, lymphocyte subpopulation levels, and therapeutic efficacy | The first and second treatment cycle: 0, 2, 6, 24, 48, 72 hours after dosing on the first day, 0 hours on the 15th day;The first treatment cycle: 0 hours on the 8th day;0 hours on the 22th day;The third and fourth treatment cycle: 0 hours on the 1st day.
  Pharmacodynamic indicators：The levels of peripheral blood serum cytokines (IL-2, IL-6, IL-8, IL-10, Interferon gamma (IFN - γ), tumor necrosis factor-α (TNF - α), interleukin 2 receptor alpha (IL-2R α), interleukin 2 receptor beta (IL-2R β), IL-2R γ, lymphocyte subsets, T cell activation markers (percentage of Cluster of (Differentiation) 25+T cells, percentage of Ki67+T cells), and the expression levels of Programmed cell death 1 (PD-1), T-cell immunoglobulin and mucin domain 3 (TIM-3), Lymphocyte-activation gene 3 (LAG-3), cytotoxic T-lymphocyte associated protein 4 (CTLA-4) on the surface of T cells.
Immunogenicity analysis- positive anti drug antibodies (ADA) | The first, third, sixth, twelfth treatment cycle: 0 hours on the first day;and End of Treatment Visit (EOT)
  Describe the number, proportion, and 95% confidence interval of positive anti drug antibodies (ADA) after medication, as well as the time and titer of ADA production
Overall response rate (ORR) | Up to 18 months
  Proportion of subjects with best response as PR, VGPR, CR, sCR.
Very good partial response rate (VGPR) | Up to 18 months
  Proportion of subjects whose best response is VGPR, CR, sCR
Complete Response (CR) | Up to 18 months
  Proportion of subjects whose best response is CR.
Strict Complete Response (sCR) Rate | Up to 18 months
  Proportion of subjects whose best response is sCR.
Negative rate of minimal residual disease (MRD) | Up to 18 months
  The proportion of subjects with negative MRD (<10-5, multicolor flow cytometry or next-generation sequencing) at any time point from the first administration of the trial drug to disease progression or before receiving new anti-tumor therapy.
Duration of remission (DOR) | Up to 18 months
  For all subjects whose best response was PR, VGPR, CR, sCR, the time from the date of first achieving PR, VGPR, CR, sCR to the date of first definite disease progression or (any cause) death(whichever occurs first).
Time to first remission (TTR) | Up to 18 months
  Among all the subjects whose best response is PR, VGPR, CR, sCR, the time from the first administration of the test drug to the date of the first PR and above remission.
Progression-free survival (PFS) | Up to 18 months
  The time between the first dose of the trial drug and the date of first definite disease progression or death (from any cause), whichever occurs first.
Overall survival (OS) | Up to 18 months
  Time from first dose of study drug to date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - West China hospital, Sichuan university, Chengdu, Sichuan